CLINICAL TRIAL: NCT00692965
Title: Sleep Quality and Presence of Sleep Disordered Breathing In An Inner City African American HIV Infected Population Aged 50 Years and Older
Brief Title: Sleep Quality and Presence of Sleep Disordered Breathing
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: J-51-2008
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: HIV Infections; Sleep
Keywords: HIV; Sleep Quality; Sleep apnea; Berlin Questionnaire; Pittsburgh Sleep Quality Index
MeSH Terms: conditions — HIV Infections; Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of our study is to survey the quality of sleep and sleep disordered breathing in a HIV infected inner city ambulatory African-American Population aged 50 years and older.

Hypothesis: African-American HIV infected individuals aged 50 years and older have a high prevalence of sleep disorders and lower quality of sleep.

DETAILED DESCRIPTION:
The purpose of our study is to survey the quality of sleep and sleep disordered breathing in a HIV infected inner city ambulatory African-American Population aged 50 years and older. A secondary objective is to investigate possible relationships between sleep quality and aspects of a patient's medical history including BMI, CD4 count, HIV viral load, history of substance abuse, psychiatric disorders, concurrent medical conditions, current HIV medications and HIV medication compliance.

Hypothesis: African-American HIV infected individuals aged 50 years and older have a high prevalence of sleep disorders and lower quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Aged 50 years and older
* HIV infected
* Receiving HIV care at the Boulevard Comprehensive Care Clinic, Duval County Health Department

Exclusion Criteria:

* Patients refusing to fill out the questionnaires
* Patients less than 50 years old
* Non-African Americans
* Persons not receiving care at the Boulevard Comprehensive Care Clinic

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected, inner city ambulatory African-American population,aged 50 years and older
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The purpose of our study is to survey the quality of sleep and sleep disordered breathing in a HIV infected inner city ambulatory African-American Population aged 50 years and older. | 10-20 minutes to complete surveys

SECONDARY OUTCOMES:
Investigate possible relationships between sleep quality and aspects of a patient's medical history | a single chart review

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Mannepalli, MD, Principal Investigator — University of Florida; Akram Khan, MD, Principal Investigator — University of Florida

REFERENCES:
- [Background] Rubinstein ML, Selwyn PA. High prevalence of insomnia in an outpatient population with HIV infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Nov 1;19(3):260-5. doi: 10.1097/00042560-199811010-00008. PMID 9803968
- [Background] Meissner HH, Riemer A, Santiago SM, Stein M, Goldman MD, Williams AJ. Failure of physician documentation of sleep complaints in hospitalized patients. West J Med. 1998 Sep;169(3):146-9. PMID 9771152
- [Background] Perkins DO, Leserman J, Stern RA, Baum SF, Liao D, Golden RN, Evans DL. Somatic symptoms and HIV infection: relationship to depressive symptoms and indicators of HIV disease. Am J Psychiatry. 1995 Dec;152(12):1776-81. doi: 10.1176/ajp.152.12.1776. PMID 8526245
- [Background] Cohen FL, Ferrans CE, Vizgirda V, Kunkle V, Cloninger L. Sleep in men and women infected with human immunodeficiency virus. Holist Nurs Pract. 1996 Jul;10(4):33-43. doi: 10.1097/00004650-199607000-00007. PMID 8717996
- [Background] Nokes KM, Kendrew J. Sleep quality in people with HIV disease. J Assoc Nurses AIDS Care. 1996 May-Jun;7(3):43-50. doi: 10.1016/S1055-3290(96)80076-8. PMID 8816356
- [Background] Norman SE, Chediak AD, Kiel M, Cohn MA. Sleep disturbances in HIV-infected homosexual men. AIDS. 1990 Aug;4(8):775-81. doi: 10.1097/00002030-199008000-00009. PMID 2261133
- [Background] Robbins JL, Phillips KD, Dudgeon WD, Hand GA. Physiological and psychological correlates of sleep in HIV infection. Clin Nurs Res. 2004 Feb;13(1):33-52. doi: 10.1177/1054773803259655. PMID 14768766
- [Background] Phillips KD, Sowell RL, Boyd M, Dudgeon WD, Hand GA; Mind-Body Research Group. Sleep quality and health-related quality of life in HIV-infected African-American women of childbearing age. Qual Life Res. 2005 May;14(4):959-70. doi: 10.1007/s11136-004-2574-0. PMID 16041893
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Reid S, Dwyer J. Insomnia in HIV infection: a systematic review of prevalence, correlates, and management. Psychosom Med. 2005 Mar-Apr;67(2):260-9. doi: 10.1097/01.psy.0000151771.46127.df. PMID 15784792
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956